CLINICAL TRIAL: NCT04508725
Title: Early Therapeutic Monitoring of Response to Therapy With Serial Ultrasound in Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Serial Ultrasound in Metastatic Renal Cell Carcinoma (mRCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alice Fan, Assistant Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-55742; RENAL0042 (Other: OnCore); NCI-2021-02327 (Registry Identifier: CTRP); 1R03CA25277601 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2020-07-29; First posted 2020-08-11 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Ultrasonography, Doppler; Receptor Protein-Tyrosine Kinases; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI) (Active Comparator): Patients are planned to be treated with vascular endothelial growth factor 2 (VEGFR2) tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI)
  Interventions: Diagnostic Test: Doppler Ultrasound; Device: SIEMENS S3000 and Verasonics Vantage 256; Drug: Standard-of-care Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI)
- Non-ICI therapy (Active Comparator): Patients are planned to be treated with non-ICI therapy
  Interventions: Diagnostic Test: Doppler Ultrasound; Device: SIEMENS S3000 and Verasonics Vantage 256; Drug: Standard-of-care non-immune checkpoint inhibitor (ICI) such as single-agent VEGFR2 TKI

INTERVENTIONS:
Diagnostic Test: Doppler Ultrasound — Power Doppler measurements will be made
Device: SIEMENS S3000 and Verasonics Vantage 256 — Vantage 256 used for power Doppler ultrasound, manufactured by Verasonics
Drug: Standard-of-care Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI) — Standard-of-care Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI).
  Other Names: VEGFR2; TKI; ICI
  Arms: Tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI)
Drug: Standard-of-care non-immune checkpoint inhibitor (ICI) such as single-agent VEGFR2 TKI — Standard-of-care non-immune checkpoint inhibitor (ICI) such as single-agent VEGFR2 TKI
  Arms: Non-ICI therapy

SUMMARY:
To assess whether changes in quantitative tumor perfusion parameters after 3 or 6 weeks of treatment, as measured by power Doppler ultrasound, can predict initial objective response, defined by current standard-of-care, to therapy at 12 weeks after start of treatment

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Pathology-confirmed diagnosis of Renal cell carcinoma (RCC)
* At least one tumor lesion greater than 1 cm in diameter, amenable to ultrasound imaging
* Written informed consent.

Specific inclusion criteria:

* Arm 1: planned to be treated with combination of VEGFR2 tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI)
* Arm 2: planned to be treated with non-ICI therapy

Exclusion Criteria:

-Any comorbid condition that, in the opinion of the treating provider or the Protocol Directors, compromises the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice C Fan, MD, Principal Investigator — Stanford University; Jeremy Dahl, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 22 participants were enrolled in the study. Twelve participants started in Arm 1 and five participants started in Arm 2. Additional two participants consecutively participated in both arms; these participants are reported in Arm 3.
  Three participants were enrolled but did not start treatment and are not included in any arm.
Groups:
- ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI): Patients were treated with vascular endothelial growth factor 2 (VEGFR2) tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI).
- ARM 2: Non-ICI Therapy: Patients were treated with non-ICI therapy.
- ARM 3: Enrolled Consecutively in Both Arms: Patients were enrolled consecutively in both arms.
Period: Overall Study
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy | ARM 3: Enrolled Consecutively in Both Arms
Started | 12 | 5 | 2
Completed | 10 | 5 | 2
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI): Patients are planned to be treated with vascular endothelial growth factor 2 (VEGFR2) tyrosine kinase inhibitor (TKI) plus immune checkpoint inhibitor (ICI)
  Doppler Ultrasound: Power Doppler measurements will be made.
  SIEMENS S3000 and Verasonics Vantage 256: Vantage 256 used for power Doppler ultrasound, manufactured by Verasonics.
- ARM 2: Non-ICI Therapy: Patients are planned to be treated with non-ICI therapy
  Doppler Ultrasound: Power Doppler measurements will be made.
  SIEMENS S3000 and Verasonics Vantage 256: Vantage 256 used for power Doppler ultrasound, manufactured by Verasonics.
- Total: Total of all reporting groups
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy | ARM 3: Enrolled Consecutively in Both Arms | Total
Number analyzed (Participants) | 12 | 5 | 2 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 1 | 2 | 12
  >=65 years | 3 | 4 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 11 | 4 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 7
  Not Hispanic or Latino | 8 | 4 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 3 | 1 | 10
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 5 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Initial Objective Response- First Participation
Description: Initial objective response was defined as having either Complete Response (CR) or Partial Response (PR) per RECIST v1.1 at first on-treatment response evaluation 8-16 weeks after initiating treatment.
Time Frame: 12 weeks
Population: Two of fourteen participants in Arm 1 were not evaluable because they were removed from the study during active participation without undergoing any response evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- ARM 2: Non-ICI Therapy: Patients were planned to be treated with non-ICI therapy.
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy
Number analyzed (Participants) | 12 | 5
Participants
  Yes (CR or PR) | 5 | 1
  No (SD or PD) | 7 | 4

2. Primary Outcome: Initial Objective Response- Second Participation
Description: Initial objective response is defined as having either Complete Response (CR) or Partial Response (PR) per RECIST v1.1 at first on-treatment response evaluation 8-16 weeks after initiating treatment.
Time Frame: 12 weeks
Population: This measure reflects outcome data from the second participation of two individuals enrolled in both Arm 1 and Arm 2. For their second participation, these individuals are grouped under Arm 3. Each participant is counted once in this outcome based on the second treatment period. For one of the two participants the outcome measure was not defined for their second treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- ARM 3: Enrolled Consecutively in Both Arms: Patients were consecutively enrolled in both study arms.
Arm/Group | ARM 3: Enrolled Consecutively in Both Arms
Number analyzed (Participants) | 1
Participants
  Yes (CR or PR) | 0
  No (SD or PD) | 1

3. Secondary Outcome: Initial Relative Change in Tumor Burden Compared to Baseline - First Participation
Description: Tumor burden was assessed as the sum of all tumor diameters at baseline compared to the first on-treatment response evaluation (8-16 weeks after the start of treatment) using RECIST v1.1 criteria
Time Frame: 8-16 weeks after the start of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy
Number analyzed (Participants) | 12 | 5
Percentage change from baseline | -16.0 (70.3) | 43.7 (94.8)

4. Secondary Outcome: Initial Relative Change in Tumor Burden Compared to Baseline - Second Participation
Description: as for outcome 3
Time Frame: 8-16 weeks after the start of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | ARM 3: Enrolled Consecutively in Both Arms
Number analyzed (Participants) | 1
Percentage change from baseline | -20.7 (0)

5. Secondary Outcome: Initial Per-Lesion Response Compared To Baseline - First Participation
Description: The relative change in tumor diameter of a single lesion between treatment 'baseline' and the first on-treatment response evaluation 8-16 weeks after the start of treatment, using RECIST v1.1 for tumor diameter measurements. This was measured as percent change and reported as mean ± standard deviation.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Units Other Than Participants: lesions
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy
Number analyzed (Participants) | 12 | 5
Number analyzed (lesions) | 18 | 5
Percentage change from baseline | -28.0 (23.0) | -4.6 (19.0)

6. Secondary Outcome: Initial Per-Lesion Response Compared To Baseline - Second Participation
Description: as for outcome 5
Time Frame: 12 weeks
Population: The total number of participants analyzed for this outcome measure reflects only those who were evaluable. Two participants in Arm 1 were not evaluable because they were removed from the study during active participation without undergoing any response evaluation. One participant in Arm 3 received a treatment during the second participation, for which the outcome measure was not defined.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Units Other Than Participants: lesions
Arm/Group | ARM 3: Enrolled Consecutively in Both Arms
Number analyzed (Participants) | 2
Number analyzed (lesions) | 2
Percentage change from baseline | -6.3 (18.7)

7. Secondary Outcome: 12-month Progression Free Survival (PFS)- First Participation
Description: PFS was defined as not having experienced any progressive disease (PD) per RECIST v1.1 within the first 12 months after initiating treatment (day 1 will be treatment start date).
Time Frame: 12 months
Population: Three of fourteen patients in arm 1 were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy
Number analyzed (Participants) | 11 | 5
Participants
  Yes (No PD and no death experienced) | 7 | 3
  No (PD or death experienced) | 4 | 2

8. Secondary Outcome: 12-month Progression Free Survival (PFS)- Second Participation
Description: PFS is defined as not having experienced any progressive disease (PD) per RECIST v1.1 within the first 12 months after initiating treatment (day 1 will be treatment start date), as a number and proportion without dispersion.
Time Frame: 12 months
Population: This outcome measure reflects 12-month progression-free survival for two participants who enrolled a second time after initial treatment. These participants are grouped under Arm 3, and each is counted once based on survival status from their second participation. For one participant the outcome measure was not defined for their second participation.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM 3: Enrolled Consecutively in Both Arms
Number analyzed (Participants) | 1
Participants
  Yes (No PD and no death experienced) | 0
  No (PD or death experienced) | 1

ADVERSE EVENTS:
Time Frame: First study ultrasound exam through 12 weeks after starting treatment.
Description: Only Adverse Events were recorded for this study that were definitely, probably, or possibly related to study procedures.
Arm/Group | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) | ARM 2: Non-ICI Therapy | ARM 3: Enrolled Consecutively in Both Arms
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 2/12 | 0/5 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1: Tyrosine Kinase Inhibitor (TKI) Plus Immune Checkpoint Inhibitor (ICI) (N=12) | ARM 2: Non-ICI Therapy (N=5) | ARM 3: Enrolled Consecutively in Both Arms (N=2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04508725/Prot_001.pdf